CLINICAL TRIAL: NCT06991972
Title: Puncture to Repigment: A Comparative Analysis Of Needling vs. Microneedling Along With NBUVB in Treatment of Non-Segmental Vitiligo
Brief Title: Comparison of Needling and Microneedling Plus Phototherapy in Localized Vitiligo Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Khyber Teaching Hospital (Other)
Responsible Party: Principal Investigator, Huma Gul, DOCTOR, Khyber Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 187/DME/KMC
Record Dates: First submitted 2025-05-19; First posted 2025-05-28 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Vitiligo; Non-segmental Vitiligo
Keywords: vitiligo; needling; microneedling
MeSH Terms: conditions — Vitiligo | interventions — Percutaneous Collagen Induction

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Needling + NBUVB(Group A) (Active Comparator)
  Interventions: Procedure: Microneedling + NBUVB
- Microneedling + NBUVB(Group B) (Active Comparator)
  Interventions: Procedure: Needling + NBUVB

INTERVENTIONS:
Procedure: Needling + NBUVB — Participants in this arm will undergo needling using a sterile 30G (4mm) needle to manually puncture and implant melanocytes from perilesional pigmented skin into depigmented lesions. The procedure will be performed once every four weeks for a total of six sessions.
  Arms: Microneedling + NBUVB(Group B)
Procedure: Microneedling + NBUVB — Participants in this arm will undergo microneedling using a Dermapen device with 1.5 mm needles to create controlled micro-injuries in depigmented skin to enhance melanocyte migration and repigmentation. This procedure will be performed once every four weeks for six sessions.
  Arms: Needling + NBUVB(Group A)

SUMMARY:
This randomized controlled trial aims to compare the efficacy of needling versus microneedling, both followed by narrowband UVB therapy, in achieving repigmentation in patients with localized stable non-segmental vitiligo.

DETAILED DESCRIPTION:
The study will enroll 80 patients aged 15-60 years with localized stable vitiligo. Participants will be randomized into two groups: one receiving needling and the other microneedling, each followed by NBUVB therapy. The primary outcome is the percentage of repigmentation at 12 weeks, assessed through digital planimetry and standardized clinical photography. Secondary outcomes include adverse effects such as erythema, post-inflammatory hyperpigmentation, infection, and scarring.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female
* Age 15-60 years
* Patients having vitiligo for more than 1 year

Exclusion Criteria:

* Patients with tendency of keloid formation or hypertrophic scarring
* Patients with any bleeding disorder, coagulation defect or using anti platelets
* Any local infection at the treatment site
* Patients who had received systemic therapy in last 6 months

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Treatment efficacy | 12 weeks
  Efficacy will be assessed at 12 weeks using the Physician's Global Assessment Scale. Improvement is defined as ≥25% repigmentation of vitiliginous patches, measured via digital planimetry and standardized clinical photography. The higher the score, the more effective is the treatment modality.
  0-25% re pigmentation= Mildimprovement 25-50% re pigmentation= Moderate improvement 51-75% re pigmentation= Good 76-100% re pigmentation= Excellent to complete

SECONDARY OUTCOMES:
Adverse effects | 12 weeks
  erythema, post-inflammatory hyperpigmentation, infection, scarring

CONTACTS AND LOCATIONS:
Overall Officials: Huma Gul Doctor, MBBS, Principal Investigator — Khyber Teaching Hospital
Locations (1):
- Khyber Teaching Hospital, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No
Patient's confidentiality may not be breached